CLINICAL TRIAL: NCT02460276
Title: A Phase II Trial of Ibrutinib, Lenalidomide and Rituximab for Patients With Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: A Trial of Ibrutinib, Lenalidomide and Rituximab for Patients With Relapsed/Refractory Mantle Cell Lymphoma
Acronym: PHILEMON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Collaborators: Celgene (Industry); Janssen, LP (Industry); Nordic Lymphoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG-MCL6
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Relapsed/Refractory Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Relapsed mantle cell lymphoma; Lenalidomide; Rituximab; Ibrutinib; Response duration; Complete remission rate; Quality of life; Overall survival; Safety
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Lenalidomide; ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide, ibrutinib and rituximab. (Experimental)
  Interventions: Drug: Lenalidomide; Drug: Ibrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide
Drug: Ibrutinib
Drug: Rituximab

SUMMARY:
In this trial, patients with mantle cell lymphoma will be included, treatment with lenalidomide, rituximab and ibrutinib will be administered in an induction phase for up to 12 cycles, cycle length 28 days. Patients with complete remission, partial response or stable disease will enter a maintenance phase with treatment with ibrutinib and rituximab until progression of disease.

The primary objective is to evaluate overall response rate, based on PET and CT.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Histologically confirmed (according to the WHO 2008, and upcoming 2015 classification) mantle cell lymphoma stage II-IV
* Received at least 1 prior rituximab-containing chemotherapy regimen
* Documented relapse or disease progression following the last anti-mantle cell lymphoma treatment
* At least 1 measurable site of disease (over 1.5 cm long axis)
* WHO performance status 0-3
* Written informed concent
* Female subjects of childbearing potential must:

  1. Understand that the study medication is expected to have a teratogenic effect
  2. Agree to use, and be able to comply with, highly effective contraception without interruption, 4 weeks Before start study drug, throughout study drug therapy (including dose interruptions) and for 12 months after the end of study drug therapy, even if she has amenorrhoea
  3. Women of childbearing potential must have a negative serum (beta-human ionic gonadotropin or urine pregnancy test at screening. Women who are pregnant or breastfeeding are ineligible for this study
* Male subjects must:

  1. Agree to use condoms throughout study drug therapy, during any dose interruption and for 3 months after cessation of study therapy if their partner is of childbearing potential and has no contraception
  2. Agree not to donate semen during study drug therapy and for 3 months after end of study drug therapy
* All subjects must agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy
* All subjects must agree not to share study medication with another person and to return all unused study drug to the investigator
* Absolute neutrophil Count (ANC) ≥ 1000/mm3
* Platelets ≥ 100,000/mm3 or ≥50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
* Alanine aminotransferase (ALT) and aspartate aminotransferase ≤ 3 x upper limit of normal (ULN).
* Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockcroft-Gault) ≥ 40 mL/min/1.73 m2
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks, therapeutic antibodies within 4 weeks, radioimmunotherapy within 10 weeks, or major surgery within 4 weeks of inclusion
* Known central nervous system lymphoma
* Other active malignancy
* Psychiatric illness or condition which could interfere with the subjects' ability to understand the requirements of the study
* Requirement of corticosteroid therapy at a dose > 10 mg prednisolone/day
* Major surgery within 4 weeks of inclusion
* History of stroke or intracranial hemorrhage within 6 months prior to inclusion
* Requirement of anticoagulation treatment with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon)
* Requirement of treatment with strong or moderate CYP3A inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Vaccination with live, attenuated vaccines within 4 weeks of inclusion
* Known history of human immunodeficiency virus (HIV) or Active hepatitis C Virus or Active Hepatitis B Virus infection or any uncontrolled Active systemic infection requiring intravenous antibiotics
* Any Life-threatening illness, Medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules or lenalidomide tablets, or put the study outcomes at undue risk
* Known hypersensitivity or allergy to rituximab, lenalidomide or ibrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate. | Change of tumor burden meassured from baseline during treatment of maximum 144 weeks.
  Tumor evaluation will be performed with CT/PET for maximum 144 weeks. Discontinuation of evaluation if the patient develops progressive disease.

CONTACTS AND LOCATIONS:
Locations (5):
- Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- Norwegian Radium Hospital, Oslo, Norway
- Sweden (2):
  - Lund University Hospital, Lund
  - Uppsala Akademiska Hospital, Uppsala

REFERENCES:
- [Derived] Jerkeman M, Eskelund CW, Hutchings M, Raty R, Wader KF, Laurell A, Toldbod H, Pedersen LB, Niemann CU, Dahl C, Kuitunen H, Geisler CH, Gronbaek K, Kolstad A. Ibrutinib, lenalidomide, and rituximab in relapsed or refractory mantle cell lymphoma (PHILEMON): a multicentre, open-label, single-arm, phase 2 trial. Lancet Haematol. 2018 Mar;5(3):e109-e116. doi: 10.1016/S2352-3026(18)30018-8. Epub 2018 Jan 29. PMID 29396091